CLINICAL TRIAL: NCT03858023
Title: Therapeutic Effects of Hippotherapy in Children With Prader-Willi Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-07-058-005
Record Dates: First submitted 2016-08-26; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Prader-Willi Syndrome
Keywords: hippotherapy; gross motor; balance; behavior
MeSH Terms: conditions — Prader-Willi Syndrome; Behavior | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hippotherapy (Experimental): Children in hippotherapy arm will participate in hippotherapy (30 min/sessions, twice a week, 15 weeks)
  Interventions: Other: Hippotherapy
- Control (No Intervention): Children in control group will not receive hippotherapy

INTERVENTIONS:
Other: Hippotherapy — The hippotherapy program consists of 2 sessions per week for 15 weeks. One session is 30-minute session. The program involves 2 therapists and 3 personnel for safety issues.
  Arms: Hippotherapy

SUMMARY:
This study evaluates the therapeutic effects of hippotherapy in children with Prader-Willi syndrome. Half of children will participate in hippotherapy for 15 weeks (30 minutes per sessions, twice a week, total 30 sessions, private lesson), while the other half will not receive hippotherapy.

DETAILED DESCRIPTION:
This study evaluates the therapeutic effects of hippotherapy in children with Prader-Willi syndrome. Half of children will participate in hippotherapy for 15 weeks (30 minutes per sessions, twice a week, total 30 sessions, private lesson), while the other half will not receive hippotherapy.

The primary purpose of this study is to investigate effect of hippotherapy on motor function of Prader-Willi syndrome patients.

The secondary purpose is to compare motor function, obesity, and behavior of the children after the intervention with those parameters before the intervention.

ELIGIBILITY:
Inclusion Criteria:

* can sit upright on the static surface
* can follow one step command

Exclusion Criteria:

* body wight > 35 kg
* serious medical conditions such as cardiac disease, pulmonary disease, uncontrolled epilepsy
* visual impairment, hearing impairment
* bleeding tendency, anticoagulation
* fracture within 6 months, major orthopedic surgery within 1 year

Ages: 42 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Clinical global Impression-Severity of illness (CGI-S) score | 15 weeks
  The Clinical Global Impression (CGI) rating scales are measures of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders. The two components of CGI were used in this study: Severity of Illness (CGI-S) and Global improvement (CGI-I). The clinician rates CGI-S on a 7-point scale from 1(normal) to 7(extremely ill) Thus, higher score means more severity outcomes
Clinical global Impression-Improvement (CGI-I) score | 15 weeks
  The clinician rates CGI-I on a 7-point scale from 1(very much improved) to 7(very much worse) respectively. Thus, higher score means worse outcomes.

SECONDARY OUTCOMES:
Gross motor function assessed by GMFM-88 (Gross Motor Function Measure) score | 15 weeks
  The 88 items of the GMFM are measured by observation of the child and scored on a 4-point ordinal scale (0=does not initiate, 1=initiates <10% of activity, 2=partially completes 10% to <100% of activity, 3=completes activity). The items are weighted equally and grouped into 5 dimensions: (1) lying and rolling (17 items), (2) sitting (20 items), (3) crawling and kneeling (14 items), (4) standing (13 items), and (5) walking, running, jumping (24 items).
Pediatric Balance Scale | 15 weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points.
PWS (Prader-Willi syndrome) hyperphagia questionnaire | 15 weeks
  The Hyperphagia Questionnaire is a robust tool for relating breakthroughs in the neurobiology of hyperphagia to in vivo food-seeking behavior and for examining the psychological and developmental correlates of hyperphagia in PWS. It has 13 items and rated on a five-point scale (1 = not a problem to 5 = severe and/or frequent problem)
Child Behavior Checklist (CBCL) | 15 weeks
  The Child Behavior Checklist (CBCL) is a widely used caregiver report form identifying problem behavior in children. CBCL asks caregivers to rate 112 problems on a three-point scale (0 not true, 1 somewhat true, 2 very true). It provides an internalizing and externalizing domain.
Obesity measured by DEXA (Dual-energy X-ray Absorptiometry) | 15 weeks
  Dual-energy X-ray Absorptiometry is a means of measuring bone mineral density (BMD). Two X-ray beams, with different energy levels, are aimed at the patient's bones. When soft tissue absorption is subtracted out, the BMD can be determined from the absorption of each beam by bone. Dual-energy X-ray absorptiometry is the most widely used and most thoroughly studied bone density measurement technology.

CONTACTS AND LOCATIONS:
Overall Officials: JEONG-YI KWON, MD, PHD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No